CLINICAL TRIAL: NCT07317609
Title: Safety and Feasibility of Neoadjuvant Immunotherapy Combined With Chemotherapy Sequenced With Endoscopic Resection for Esophageal Cancer (Endosurgery-02)
Brief Title: Neoadjuvant Immunotherapy Combined With Chemotherapy Sequenced With Endoscopic Resection for Esophageal Cancer (Endosurgery-02)
Acronym: Endosurgery-02
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiZhongshanEndosurgery02
Record Dates: First submitted 2025-11-25; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: neoadjuvant, chemoimmunotherapy, tislelizumab, carboplatin, nab-paclitaxel, endoscopic submucosal dissection/ESD
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — tislelizumab; Carboplatin; 130-nm albumin-bound paclitaxel; Endoscopic Mucosal Resection; Esophagectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Tislelizumab + Carboplatin + Nab-Paclitaxel (Experimental): Participants receive neoadjuvant chemoimmunotherapy for at least two 3-week cycles: tislelizumab 200 mg IV on Day 1 (Q3W) plus carboplatin AUC 3-5 IV on Day 1 (Q3W) and nab-paclitaxel ≤260 mg/m² IV on Day 1 (Q3W; ~30-minute infusion). Safety is assessed during treatment. About 3-4 weeks after completing ≥2 cycles, participants undergo clinical reassessment (physical exam, labs, and imaging including endoscopy/EUS and PET/CT or CT of neck, chest, and upper abdomen) and tumor response is evaluated by RECIST 1.1. If clinical complete response (cCR) is achieved without obvious nodal disease, endoscopic resection is performed 3-6 weeks after neoadjuvant therapy; otherwise, patients proceed to standard esophagectomy or concurrent chemoradiation per investigator judgment.
  Interventions: Drug: Tislelizumab; Drug: Carboplatin; Drug: Nab-paclitaxel; Procedure: Endoscopic resection; Procedure: Esophagectomy; Radiation: Concurrent chemoradiation

INTERVENTIONS:
Drug: Tislelizumab — Fixed-dose anti-PD-1 monoclonal antibody 200 mg IV on Day 1 of each 3-week cycle (Q3W) as neoadjuvant therapy, administered before any local resection. Given for ≥2 cycles unless contraindicated. Used in combination with carboplatin and nab-paclitaxel in a single-arm regimen; no placebo or comparator.
Drug: Carboplatin — Intervention Description: AUC 3-5 IV on Day 1, Q3W, for ≥2 cycles in combination with tislelizumab and nab-paclitaxel as neoadjuvant therapy.
Drug: Nab-paclitaxel — ≤260 mg/m² IV on Day 1, Q3W (~30-min infusion) for ≥2 cycles, combined with tislelizumab and carboplatin in the neoadjuvant regimen.
Procedure: Endoscopic resection — Endoscopic resection (e.g., ESD/EFTR) performed 3-6 weeks after completing ≥2 neoadjuvant cycles only if clinical complete response (cCR) is achieved without clear nodal metastasis, based on endoscopy/EUS and imaging. Technique follows institutional standards with curative intent and margin assessment.
Procedure: Esophagectomy — Standard surgical esophagectomy (McKeown/Ivor-Lewis procedures) for participants not meeting cCR criteria or deemed unsuitable for endoscopic resection after reassessment. Conducted per institutional standard of care, with lymphadenectomy as appropriate.
Radiation: Concurrent chemoradiation — Concurrent chemoradiation per institutional standard for participants not eligible for endoscopic resection and managed non-surgically after reassessment. External-beam radiation delivered with concurrent platinum-taxane chemotherapy as clinically indicated; specific dose/fractionation per treating radiation oncologist.

SUMMARY:
This single-center, prospective, single-arm study will evaluate whether giving neoadjuvant chemoimmunotherapy can safely shrink esophageal cancer and allow organ-preserving endoscopic removal in selected patients. Adults with esophageal cancer will receive at least two 3-week cycles of a PD-1 inhibitor (tislelizumab 200 mg on Day 1) plus carboplatin (AUC 3-5, Day 1) and nab-paclitaxel (≤260 mg/m², Day 1). During treatment, routine safety tests are performed. About 3-4 weeks after completing at least two cycles, participants undergo clinical reassessment with examinations and imaging (such as endoscopy, endoscopic ultrasound, PET/CT or CT of the neck, chest, and upper abdomen) to evaluate tumor shrinkage and possible spread. Tumor response is assessed using RECIST 1.1. If a clinical complete response is achieved without obvious nodal disease, endoscopic resection may be performed to preserve the esophagus; otherwise, patients may proceed to surgery or concurrent chemoradiation per clinical judgment. The study focuses on feasibility and safety of this organ-preserving approach and describes tumor responses after therapy. Potential benefits include tumor shrinkage and avoiding major surgery in selected cases; risks include side effects of standard chemotherapy/immunotherapy and procedure-related discomforts from biopsies or endoscopic treatments.

ELIGIBILITY:
Cohort A - Potentially resectable ESCC:

Inclusion Criteria：

1. Age range: 18-80 years old;
2. Patients diagnosed with esophageal squamous cell carcinoma (ESCC) through histopathological examination of biopsy tissues from the primary tumor;
3. Patients with potentially resectable esophageal cancer confirmed by imaging and endoscopic examinations (T1b-3, N0, M0, with a tumor size not exceeding 5 cm and occupying less than 2/3 of the luminal circumference); Patients who have not received any antitumor treatment, including but not limited to surgery, radiotherapy, chemotherapy, immunotherapy, and targeted therapy;
4. Patients with a preoperative Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
5. Patients with a preoperative American Society of Anesthesiologists (ASA) physical status classification of I-III;
6. Female patients of reproductive age should have a negative pregnancy test and be willing to use effective contraceptive methods during the study period;
7. Patients who have signed the informed consent form.

Exclusion Criteria:

1. Patients with potential tracheoesophageal fistula or aortoesophageal fistula;
2. Patients with severe malnutrition or requiring tube feeding;
3. Patients with other malignancies that have not been cured within the past 2 years (except for cured basal cell carcinoma of the skin and cured carcinoma in situ of the cervix);
4. Patients with active autoimmune diseases or a history of autoimmune diseases or symptoms that require systemic corticosteroid treatment or anti-autoimmune drug therapy;
5. Immunocompromised patients, or patients who are still receiving systemic steroids (prednisone > 10 mg/day or equivalent) or other forms of immunosuppressive therapy within 7 days before the first dose of neoadjuvant therapy in this study;
6. Patients with active infections requiring systemic treatment within 7 days before the first neoadjuvant therapy in this study;
7. Patients with a history of allogeneic organ or stem cell transplantation;
8. Patients with allergies to drugs or related components involved in this study;
9. Patients who are currently participating in any other clinical study.

Cohort B - Surgery-contraindicated ESCC:

Inclusion Criteria:

1. Individuals aged above 18 years;
2. Patients diagnosed with esophageal squamous cell carcinoma through histopathological examination of biopsy tissues from the primary tumor;
3. Patients with esophageal cancer deemed as surgically contraindicated (including those with cervical esophageal cancer, surgical contraindications, those who refuse surgery, or those considered high-risk for esophagectomy, defined as having at least one of the following characteristics: (1) age over 75 years, (2) Charlson comorbidity index >= 2, (3) presence of moderate lung dysfunction, (4) malnutrition (with a body mass index below 18 kg/m^2)), with a clinical staging of cT1b-3N0M0, a tumor size not exceeding 5 cm, and occupying less than 2/3 of the luminal circumference;
4. Patients who have not undergone any antitumor treatment, including but not limited to surgery, radiotherapy, chemotherapy, immunotherapy, and targeted therapy;
5. Female patients of reproductive age should have a negative pregnancy test and be willing to adopt effective contraceptive measures during the study period;
6. Patients who have signed the informed consent form.

Exclusion Criteria:

1. Patients with allergies to the drugs or related components involved in this study;
2. Patients who are currently participating in any other clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Organ preservation rate | Up to 12 months after completion of neoadjuvant therapy
  Proportion of enrolled participants who achieve esophageal organ preservation after neoadjuvant therapy, defined as: (1) clinical complete response at reassessment ~3-4 weeks after ≥2 cycles; (2) endoscopic tumor resection (e.g., ESD) performed 3-6 weeks after therapy with curative intent and negative margins (R0) when resection is undertaken; and (3) no planned or salvage esophagectomy through 12 months. Participants who require esophagectomy, have persistent/progressive disease precluding endoscopic therapy, or die before assessment are counted as non-preserved.
Overall safety: incidence of Grade ≥3 adverse events related to drug, endoscopic procedures, surgery, or radiation | Adverse event was assessed peri-procedural of drug-using, endoscopic procedures, surgery, or radiation up to 30 days
  Proportion of participants with at least one Grade ≥3 adverse event from any study-specified modality:
  1. Drug-related treatment-related adverse events (TRAEs) graded by CTCAE v5.0 .
  2. Endoscopic complications when resection is performed (clinically significant bleeding requiring intervention, perforation, or stricture requiring dilation/stenting), adjudicated per institutional/ASGE criteria;
  3. Surgical morbidity after esophagectomy (Clavien-Dindo grade ≥III within 90 days of surgery);
  4. Radiation toxicities among those receiving concurrent chemoradiation (CTCAE v5.0 grade ≥3).
  Serious adverse events (SAEs) (death, life-threatening event, inpatient hospitalization/prolongation, disability, or other medically important event) and 30-/90-day all-cause mortality are captured; if multiple events occur, the worst grade counts for this composite endpoint
Two-year overall survival rate | From Day 1 of the first neoadjuvant dose to 24 months
  Proportion of participants alive 24 months after index date regardless of cause of death (all-cause mortality). The index date is Day 1 of the first neoadjuvant cycle. Survival status is ascertained from clinic visits, hospital records, and scheduled follow-up contacts. The OS rate at 24 months will be estimated using the Kaplan-Meier method with 95% confidence interval. Participants alive at last contact before 24 months are censored at that date; deaths at any time up to 24 months count as events, including those occurring after endoscopic resection, esophagectomy, or chemoradiation.
Biomarkers | Baseline and the day 1 of endoscopy or surgery
  Tumor tissue samples and blood samples will be collected for tumor biomarker analysis, including but not limited to analyses of metabolic markers, circulating tumor cells (CTCs), circulating tumor DNA (ctDNA), T-cell receptor sequencing (TCR-seq), and RNA sequencing (RNA-seq).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wu H, Leng X, Liu Q, Mao T, Jiang T, Liu Y, Li F, Cao C, Fan J, Chen L, Chen Y, Yao Q, Lu S, Liang R, Hu L, Liu M, Wan Y, Li Z, Peng J, Luo Q, Zhou H, Yin J, Xu K, Lan M, Peng X, Lan H, Li G, Han Y, Zhang X, Xiao ZJ, Lang J, Wang G, Xu C. Intratumoral Microbiota Composition Regulates Chemoimmunotherapy Response in Esophageal Squamous Cell Carcinoma. Cancer Res. 2023 Sep 15;83(18):3131-3144. doi: 10.1158/0008-5472.CAN-22-2593. PMID 37433041
- [Result] Ajani JA, D'Amico TA, Bentrem DJ, Chao J, Corvera C, Das P, Denlinger CS, Enzinger PC, Fanta P, Farjah F, Gerdes H, Gibson M, Glasgow RE, Hayman JA, Hochwald S, Hofstetter WL, Ilson DH, Jaroszewski D, Johung KL, Keswani RN, Kleinberg LR, Leong S, Ly QP, Matkowskyj KA, McNamara M, Mulcahy MF, Paluri RK, Park H, Perry KA, Pimiento J, Poultsides GA, Roses R, Strong VE, Wiesner G, Willett CG, Wright CD, McMillian NR, Pluchino LA. Esophageal and Esophagogastric Junction Cancers, Version 2.2019, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 Jul 1;17(7):855-883. doi: 10.6004/jnccn.2019.0033. PMID 31319389
- [Result] NCT02551458
- [Result] Noordman BJ, Wijnhoven BPL, Lagarde SM, Boonstra JJ, Coene PPLO, Dekker JWT, Doukas M, van der Gaast A, Heisterkamp J, Kouwenhoven EA, Nieuwenhuijzen GAP, Pierie JEN, Rosman C, van Sandick JW, van der Sangen MJC, Sosef MN, Spaander MCW, Valkema R, van der Zaag ES, Steyerberg EW, van Lanschot JJB; SANO-study group. Neoadjuvant chemoradiotherapy plus surgery versus active surveillance for oesophageal cancer: a stepped-wedge cluster randomised trial. BMC Cancer. 2018 Feb 6;18(1):142. doi: 10.1186/s12885-018-4034-1. PMID 29409469
- [Result] Zhang X, Eyck BM, Yang Y, Liu J, Chao YK, Hou MM, Hung TM, Pang Q, Yu ZT, Jiang H, Law S, Wong I, Lam KO, van der Wilk BJ, van der Gaast A, Spaander MCW, Valkema R, Lagarde SM, Wijnhoven BPL, van Lanschot JJB, Li Z. Accuracy of detecting residual disease after neoadjuvant chemoradiotherapy for esophageal squamous cell carcinoma (preSINO trial): a prospective multicenter diagnostic cohort study. BMC Cancer. 2020 Mar 6;20(1):194. doi: 10.1186/s12885-020-6669-y. PMID 32143580
- [Result] Noordman BJ, Spaander MCW, Valkema R, Wijnhoven BPL, van Berge Henegouwen MI, Shapiro J, Biermann K, van der Gaast A, van Hillegersberg R, Hulshof MCCM, Krishnadath KK, Lagarde SM, Nieuwenhuijzen GAP, Oostenbrug LE, Siersema PD, Schoon EJ, Sosef MN, Steyerberg EW, van Lanschot JJB; SANO study group. Detection of residual disease after neoadjuvant chemoradiotherapy for oesophageal cancer (preSANO): a prospective multicentre, diagnostic cohort study. Lancet Oncol. 2018 Jul;19(7):965-974. doi: 10.1016/S1470-2045(18)30201-8. Epub 2018 Jun 1. PMID 29861116
- [Result] Ge F, Huo Z, Cai X, Hu Q, Chen W, Lin G, Zhong R, You Z, Wang R, Lu Y, Wang R, Huang Q, Zhang H, Song A, Li C, Wen Y, Jiang Y, Liang H, He J, Liang W, Liu J. Evaluation of Clinical and Safety Outcomes of Neoadjuvant Immunotherapy Combined With Chemotherapy for Patients With Resectable Esophageal Cancer: A Systematic Review and Meta-analysis. JAMA Netw Open. 2022 Nov 1;5(11):e2239778. doi: 10.1001/jamanetworkopen.2022.39778. PMID 36322089
- [Result] Wang J, Zhang K, Liu T, Song Y, Hua P, Chen S, Li J, Liu Y, Zhao Y. Efficacy and safety of neoadjuvant immunotherapy combined with chemotherapy in locally advanced esophageal cancer: A meta-analysis. Front Oncol. 2022 Sep 5;12:974684. doi: 10.3389/fonc.2022.974684. eCollection 2022. PMID 36158679
- [Result] Fan M, Dai L, Yan W, Yang Y, Lin Y, Chen K. Efficacy of programmed cell death protein 1 inhibitor in resection transformation treatment of esophageal cancer. Thorac Cancer. 2021 Aug;12(15):2182-2188. doi: 10.1111/1759-7714.14054. Epub 2021 Jun 17. PMID 34137505
- [Result] Sun JM, Shen L, Shah MA, Enzinger P, Adenis A, Doi T, Kojima T, Metges JP, Li Z, Kim SB, Cho BC, Mansoor W, Li SH, Sunpaweravong P, Maqueda MA, Goekkurt E, Hara H, Antunes L, Fountzilas C, Tsuji A, Oliden VC, Liu Q, Shah S, Bhagia P, Kato K; KEYNOTE-590 Investigators. Pembrolizumab plus chemotherapy versus chemotherapy alone for first-line treatment of advanced oesophageal cancer (KEYNOTE-590): a randomised, placebo-controlled, phase 3 study. Lancet. 2021 Aug 28;398(10302):759-771. doi: 10.1016/S0140-6736(21)01234-4. PMID 34454674
- [Result] Chan KKW, Saluja R, Delos Santos K, Lien K, Shah K, Cramarossa G, Zhu X, Wong RKS. Neoadjuvant treatments for locally advanced, resectable esophageal cancer: A network meta-analysis. Int J Cancer. 2018 Jul 15;143(2):430-437. doi: 10.1002/ijc.31312. Epub 2018 Mar 8. PMID 29441562
- [Result] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Result] Medical Research Council Oesophageal Cancer Working Group. Surgical resection with or without preoperative chemotherapy in oesophageal cancer: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1727-33. doi: 10.1016/S0140-6736(02)08651-8. PMID 12049861
- [Result] Morgan E, Soerjomataram I, Rumgay H, Coleman HG, Thrift AP, Vignat J, Laversanne M, Ferlay J, Arnold M. The Global Landscape of Esophageal Squamous Cell Carcinoma and Esophageal Adenocarcinoma Incidence and Mortality in 2020 and Projections to 2040: New Estimates From GLOBOCAN 2020. Gastroenterology. 2022 Sep;163(3):649-658.e2. doi: 10.1053/j.gastro.2022.05.054. Epub 2022 Jun 4. PMID 35671803
- [Result] Sugimura K, Miyata H, Tanaka K, Makino T, Takeno A, Shiraishi O, Motoori M, Yamasaki M, Kimura Y, Hirao M, Fujitani K, Yasuda T, Mori M, Eguchi H, Yano M, Doki Y. Multicenter Randomized Phase 2 Trial Comparing Chemoradiotherapy and Docetaxel Plus 5-Fluorouracil and Cisplatin Chemotherapy as Initial Induction Therapy for Subsequent Conversion Surgery in Patients With Clinical T4b Esophageal Cancer: Short-term Results. Ann Surg. 2021 Dec 1;274(6):e465-e472. doi: 10.1097/SLA.0000000000004564. PMID 33065643
- [Result] Shapiro J, van Lanschot JJB, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch ORC, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Bilgen EJS, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS study group. Neoadjuvant chemoradiotherapy plus surgery versus surgery alone for oesophageal or junctional cancer (CROSS): long-term results of a randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1090-1098. doi: 10.1016/S1470-2045(15)00040-6. Epub 2015 Aug 5. PMID 26254683